CLINICAL TRIAL: NCT07379697
Title: The Feasibility of Measuring Unipolar Atrial Local Potentials From a Range of Pulsed Field Ablation Catheters. The MULTI PFA (EU) Study
Brief Title: Measuring Local Potentials in PFA. MULTI PFA (EU)
Acronym: MULTI PFA
Status: Not yet recruiting | Type: Observational
Sponsor: CathVision ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: CVPFA-004
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a prospective, multi-center, exploratory, observational study with the ECGenius® System and the PFAnalyzer software module in PFA cases using the Affera Sphere 9, FaraWave, PulseSelect, Volt or VariPulse PFA systems. The cohort will be adult patients with paroxysmal or persistent atrial fibrillation (AF) who undergo PVI using PFA.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrhythmia and is associated with a five-fold increase in stroke. Pulmonary vein isolation (PVI) has become a first-line treatment for paroxysmal AF. PVI is achieved by ablating cardiac tissue around the pulmonary veins. Until recently, this has been achieved using thermal energy. However, more recently a new energy source known as pulsed field ablation (PFA) has been introduced. As PFA is tissue selective, it preserves the function of nearby structures such as the esophagus and phrenic nerve making it safer to use. As PFA is delivered in short bursts of high energy, it is also more efficient and leads to shorter procedures. However, the catheters designed to deliver PFA differ to those used previously and do not provide the same information about efficacy, making it more difficult for the operator to ascertain if the lesions have successfully isolated the pulmonary vein. This exploratory observational study will assess the utility of a software module designed to measure the local potential derived from the unipolar electrogram recorded at the electrode that has delivered the PFA. During the procedure, the study will collect data only and all analysis of the output of the PFAnalyzer software module will be made off-line once the procedure is complete. The operator will follow the hospital's standard of care during the procedure, and the software module will not be used to guide therapy, nor will there be any additional time added to the procedure.

The study is a prospective, multi-center, exploratory, observational study with the ECGenius® System and the PFAnalyzer software module in PFA cases using the Affera Sphere 9, FaraWave, PulseSelect or VariPulse PFA systems. The cohort will be adult patients with paroxysmal or persistent atrial fibrillation (AF) who undergo PVI using PFA.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects undergoing first time pulmonary vein isolation indicated by investigator for the treatment of atrial fibrillation.

  2. Male or non-pregnant female aged ≥21 years. 3. Able and willing to provide written informed consent prior to any clinical investigation related procedure.

  4. Subjects in sinus rhythm at the time of the PFA application.

Exclusion Criteria:

* 1. Pregnant or nursing subjects. 2. Current participation in another investigational drug or device study that interferes with this study.

  3. Subjects who, in the opinion of the investigator, are not candidates for this study.

  4. Patients who have had a prior ablation procedure. 5. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.

  6. Life expectancy is less than 12 months, in the opinion of the investigator. 7. Subjects who, in the opinion of the investigator, are considered part of any vulnerable population.

  8. Subjects unlikely to be in sinus rhythm at the time of the procedure or unlikely to remain in sinus rhythm after cardioversion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation referred for a cardiac ablation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-04-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify a clinically meaningful threshold for residual potentials after PFA delivery | At the time of the procedure
  The peak-to-peak voltage in mV of post-PFA signals identified as local potentials by an experienced electrophysiologist will be recorded
Identify a clinically meaningful threshold for residual potentials after PFA delivery | At the time of the procedure
  The peak-to-peak voltage of local potentials identified by an experienced electrophysiologist will be measured in mV by the PFAnalyzer software